CLINICAL TRIAL: NCT05480202
Title: Effect of Thoracic Block Technique on Atelectasis in Children on Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Abdallah Amin, Scientific researcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P. T. REC/012/003483
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Atelectasis; Intensive Care Unit; Children
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic block technique and designed chest physical therapy program (Experimental): Manual compression on healthy lung for 20 seconds and rest for 20 seconds, total time 20 minutes and percussion,vibration , postural drainage one session time for 35 minutes every day for ten days
  Interventions: Other: Thoracic block technique
- Designed chest physical therapy program (Active Comparator): Percussion, vibration and postural drainage for 30 minutes every day for ten days
  Interventions: Other: Designed chest physical therapy program

INTERVENTIONS:
Other: Thoracic block technique — Manual compression of the healthy lung during expiration associated with the use of invasive or non invasive mechanical ventilation
  Other Names: Technique of insufflation to reverse atelectasis
  Arms: Thoracic block technique and designed chest physical therapy program
Other: Designed chest physical therapy program — Percussion, vibration and postural drainage
  Arms: Designed chest physical therapy program

SUMMARY:
Statement of the problem:

• Does the thoracic block technique has effect on atelectasis in Children on Mechanical Ventilation?

Null hypothesis:

• there is effect of thoracic block technique on atelectasis in children on Mechanical ventilation.

DETAILED DESCRIPTION:
Subjects:

The study targets the children from both sexes. Sample size estimation will be carried out to determine the recruited number of children, selected randomly from Cairo University pediatric specialized hospital intensive care units ,Cairo to participate in the study

Study design:

Randomized controlled clinical trial.

A. Inclusion criteria:

1. age range from 6 months to 4 years .
2. diagnosed with pneumonia, receiving Mechanical ventilation.
3. start from second day of admission to intensive care unit.
4. have unilateral mild to moderate atelectasis according to medical referral .
5. should be vitally stable during the session.

B. Exclusion criteria:

The children will be excluded from the study if they had one of the following:

1. medically unstable ( examples: tachycardia and tachypnea).
2. uncontrolled convulsion.
3. irritable or moderate to sever pain
4. rib fracture
5. pneumothorax

Children will be assessed by measuring heart rate, respiratory rate, chest x-ray, arterial blood gases,dynamic compliance, oxygen saturation index before and after ten days of receiving intervention

ELIGIBILITY:
Inclusion Criteria:

1. age range from 6 months to 4 years .
2. diagnosed with pneumonia, receiving Mechanical ventilation.
3. start from second day of admission to intensive care unit.
4. have unilateral mild to moderate atelectasis according to medical referral.
5. should be vitally stable during the session.

B. Exclusion criteria:

The children were excluded from the study if they had one of the following:

Exclusion Criteria:

The children were excluded from the study if they had one of the following:

1. medically unstable ( examples: tachycardia and tachypnea).
2. uncontrolled convulsion.
3. irritable or moderate to sever pain
4. rib fracture
5. pneumothorax

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Assessment of heart rate and respiratory rate | 10 days for each participant
  Assessment of change in heart rate and respiratory rate will be carried out by using electro cardiograph electrodes and pulse oximeter.
Assessment of atelectasis in chest x ray | 10 days for each participant
  Assessment of atelectasis in chest x ray will be carried out by comparing presence, extent and distribution of atelectasis in x ray film before and intervention
Assessment of arterial blood gases test | 10 days for each participant
  Assessment of change in arterial blood gases test will be carried out by comparing results before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Abdallah, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt